CLINICAL TRIAL: NCT07039357
Title: A Single Centre, Open-label Clinical Investigation Confirming the Safety and Accuracy of the Glyconics-DS in Assessment of Glycated Nail Keratin in Individuals With or Without Known T2DM: a Confirmatory Performance Evaluation of the Glyconics SW Package Delivering the Dichotomised Screening Test Results in a Known Population.
Brief Title: Reconfirming the Safety and Performance of the Glyconics-DS System in Known Populations With and Without Diabetes
Acronym: ANODE04
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glyconics Ltd (Industry)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NIRDM-SXCIP04
Record Dates: First submitted 2025-06-10; First posted 2025-06-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apparently healthy volunteers without known diabetes (Experimental): Both methods for assessment of glycaemia will be applied in this group as well
  Interventions: Device: Near-infrared (spectroscopy) for non-invasive assessment of glycated keratin of nail
- People with known T2DM (Experimental): Both methods for assessment of glycaemia will be applied in this group as well
  Interventions: Device: Near-infrared (spectroscopy) for non-invasive assessment of glycated keratin of nail

INTERVENTIONS:
Device: Near-infrared (spectroscopy) for non-invasive assessment of glycated keratin of nail — both interventions will be applied in both participant groups
  Other Names: HbA1c analysis by point-of-care device

SUMMARY:
A single-site, open label, confirmatory study assessing two biomarkers indicative of levels of glycaemia; glycated keratin in fingernails and glycated haemoglobin (HbA1c). Screening for diabetes

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adults (≥18 years of age) with known (n=50) or unknown T2DM status (n=50) willing to participate in and provide a written consent for the study
* willingness to undertake assisted assessment of glycaemia by both the NIR spectra measurement, and HbA1c by finger prick test
* Individuals with at least one visually assessed undamaged, intact (preferably middle) fingernail

Exclusion Criteria:

* Individuals with any known medical conditions impacting the PoC device assessment methodology for glycaemia, such as

  * Severe forms of anaemia (diagnosed iron deficiency, sickle cell anaemia or similar)
  * haemoglobinopathies or atypical haemoglobin subtypes not detectable by the assay
  * severe renal impairment (CKD stage III-IV) or decompensated hepatic disease
  * severe Vitamin D deficiency (diagnosed or measured 25(OH)D3 < 25 nmol/ml)
  * known severe immunodeficiency such as HIV, malignancy or other chronic condition significantly impacting assessment of glycaemia
  * eating disorders (as per clinical assessment)
  * recent (within 28 days) blood donation
  * known / diagnosed other diabetes such as T1DM, GDM, MODY, etc.
* For the Glyconics-DS device / targeted nail:

  * Mechanical damage or marks on the surface of the nail after removal of nail polish, or
  * Use of acrylic or gel nail decoration and polish, which cannot be removed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Specificity (%) meeting the acceptability criteria in identification correct dichotomised output / diabetes screening test result (being above or below HbA1c level of 48 mmol/mol) | 10 minutes
  Acceptance criteria for specificity is to demonstrate a result being at least or above 75%
Sensitivity (%) meeting the acceptability criteria in identification correct dichotomised output / diabetes screening test result (being above or below HbA1c level of 48 mmol/mol) | 10 minutes
  Acceptance criteria for sensitivity is to demonstrate a result being at least or above 30%

SECONDARY OUTCOMES:
Secondary performance measure and accuracy: False positive / negative rates for the screening test result | 10 minutes
  Assessment of sensitivity and specificity -derived false positive / false negative rates in % for chemometric model outcomes for HbA1c cut-off value of 48 mmol/mol (6.5%) in the study cohort n=100, in individuals with and without known T2DM.

OTHER OUTCOMES:
Patient reported outcomes: test preference | 2 minutes
  Rapid participant feedback based on preferred test methodology (Glyconics-DS vs PoC finger prick test), both cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Liver Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The plan will be completed during the incoming weeks